CLINICAL TRIAL: NCT00816192
Title: Comparison of Externally Versus Internally Cooled Tip Catheter in Achieving Long-term Electrical Isolation of Pulmonary Veins in Paroxysmal Atrial Fibrillation
Brief Title: Comparison of Externally Versus Internally Cooled Tip Catheter Ablation in Paroxysmal Atrial Fibrillation
Acronym: CATAFABL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The production of the device used in this study has been suspended.
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2008/27
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Atrial Fibrillation
Keywords: FA; Atrial fibrillation; Catheter; Ablation; RF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The externally irrigated-tip catheter is an "open system" in which saline is continuously infused and empties into the blood pool. For the externally irrigated-tip catheter, RF energy delivery settings were: power ≤ 35 watts and temperature ≤ 43°C with a variable flow-rate to obtain a temperature around 40°C.
  Interventions: Procedure: Long-term electrical isolation of pulmonary veins
- 2 (Experimental): For the internally irrigated tip catheter (reference catheter), radiofrequency (RF) energy delivery settings will be: power ≤ 35 watts, temperature ≤ 47◦C and a fixed flow rate of 0.6 ml/s.
  The advantage of the Chili thermo-cooled tip system is that no saline solution leaves the catheter system and flows into the patient.
  Interventions: Procedure: Long-term electrical isolation of pulmonary veins

INTERVENTIONS:
Procedure: Long-term electrical isolation of pulmonary veins — All AAD except amiodarone will be stopped five half-lives before the procedure. Our ablation protocol will require 3 catheters. A quadripolar stearable mapping catheter was inserted into the coronary sinus, a decapolar circular mapping catheter was placed at the antrum of the PV after transeptal puncture to help for electrical disconnection of all four PV with the randomized ablation catheter. After transseptal access, an intravenous bolus of heparin was administered and repeated 3 to 4 hours later. Atrial burst will then be used to induce AF. With the ablation catheter positioned proximal to Lasso catheter on the atrial aspect of PV ostium, isolation will be performed.

SUMMARY:
There is no study comparing safety/efficacy of externally vs internally cooled tip catheters in patients undergoing ablation for paroxysmal atrial fibrillation (pAF).

The primary objective is to compare safety and efficacy of externally irrigated-tip catheter versus internally irrigated-tip catheter in achieving long term electrical isolation (EI) of pulmonary veins (PV) in paroxysmalatrial fibrillation (pAF).

DETAILED DESCRIPTION:
Atrial fibrillation is the most common of all sustained cardiac arrhythmias, with the prevalence increasing with age to up to 5 percent in persons more than 65 years of age, to 10 percent in persons more than 80 years of age and it is a major cause of stroke.

Since its introduction into clinical practice, catheter ablation (CA) aimed at cure of atrial fibrillation (AF) has become increasingly prevalent. Different techniques have been proposed and are currently under investigation in various electrophysiology (EP) laboratories, with increasing knowledge of the pathophysiology of human AF and critical assessment of clinical outcome after the curative procedure. The favorable results reported in different studies have fueled enthusiasm for CA of AF, with the number of ablation procedures increasing from 1994 to the present time. However, these technologies have varied catheter designs, ranging from different forms of irrigation (external or internal irrigation). The increase of the rate of success of the AF by ablation with the development of new catheters has permitted a considerable reduction of the medical treatment and the disappearance of grave complications. The procedure will be " standard " with isolation of pulmonary veins and block through the cavo-tricuspid isthmus obtained.

Following completion of the procedure, patients will have anti vitamin K drug therapy for 3 months and antiarrhythmic drug for 1 month in case of early atrial arrhythmia recurrence. Two-dimensional echocardiogram will be performed systematically prior to discharge. All 3 months, long-term follow-up consisted from the date of the ablation procedure with consultation, stress test, holter-ECG (24 h) and echocardiography. At 3 months a repeat EP procedure will be performed in patients with AF recurrence to assess whether or not lines are still blocked. If not, RF will be delivered to block them again and cure AF.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Drug refractory paroxysmal AF with episods lasting <24hours
* Follow-up possible at one of the 2 institutions performing the study
* Oral agreement of the patient after reading the document of information

Exclusion Criteria:

* Pregnancy
* Psychiatric troubles not stabilized
* Contraindication to undergo AF ablation
* Previous attempt at AF ablation
* Cardioversion for AF
* No oral agreement of the patient for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
RF duration (in minutes) to succeed in PVs isolation | Along intervention

SECONDARY OUTCOMES:
The absence of pAF | at 3 and 6 months off AAD
The determination of serious adverse events (Complications resulting from vascular access will not be included in this category). | During 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel HAÏSSAGUERRE, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - University Hospital, Bordeaux
  - Clinique Pasteur, Toulouse